CLINICAL TRIAL: NCT00881478
Title: Family Intervention for Obese Children Using Portion Control Strategy (F.O.C.U.S.) for Weight Control- A Randomized Controlled Trial
Brief Title: Family Intervention for Obese Children Using Portion Control Strategy for Weight Control
Acronym: FOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Josephine Ho, Assistant Professor, Faculty of Medicine, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E22161
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2011-10

CONDITIONS: Obesity
Keywords: Obesity; Children; Dyslipidemia; Hypertension
MeSH Terms: conditions — Obesity; Dyslipidemias; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition counselling alone (Active Comparator): Nutrition counseling session with registered dietician
  Interventions: Other: Nutrition counseling
- Nutrition counselling + portion control (Experimental): Nutrition counseling with registered dietician in addition to teaching about use of a portion control tool
  Interventions: Other: Nutrition counseling + portion control tool

INTERVENTIONS:
Other: Nutrition counseling + portion control tool — Nutrition counseling with registered dietician in addition to teaching about how use of a portion control tool
  Arms: Nutrition counselling + portion control
Other: Nutrition counseling — Nutrition counseling with registered dietician
  Arms: Nutrition counselling alone

SUMMARY:
Obesity in children is a serious disease that is associated with increased mortality and decreased life expectancy. A simple tool used to assist in controlling portions (and therefore calorie intake) at mealtime would be of benefit in promoting weight maintenance and/or loss. The purpose of this study is to assess the efficacy of a family intervention using a portion control tool to help control weight in obese children. The investigators hypothesize that the use of portion control tools by the parents and child will result in a greater decrease in the child's BMI over a 6 month period compared with the control group.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to assess the efficacy of a portion control tool to help improve body mass index in obese children over a 6 months period. This study will also assess whether this weight control strategy results in improvement of blood pressure, waist circumference, and biomarkers of obesity including plasma visfatin, adiponectin, fasting lipid profile and apolipoprotein B, liver function tests and fasting insulin and glucose. Both the intervention and the control group will receive a one hour session of standard dietary counseling from a registered dietician at baseline regarding healthy eating habits, appropriate portion sizes and the Canada Food Guide. The duration of this study will be 6 months. Baseline measurements will be taken at the initial visit and again at 3 months and 6 months. Each participants' height and weight will be measured, and BMI will be calculated. Waist circumference and blood pressure will also be measured. A blood sample will be drawn at baseline and 6 months for a fasting lipid profile, fasting insulin, and glucose levels. Measurement of plasma visfatin and adiponectin levels using ELISA will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* age 8 years old to 16 years old
* BMI greater than or equal to the 85th percentile for age and gender

Exclusion Criteria:

* patients currently taking a weight loss medication
* gastrointestinal disorder
* psychiatric illness under the care of a psychiatrist
* Cushing's syndrome
* hypothalamic or genetic etiology of obesity
* uncontrolled or untreated thyroid disease
* current diagnosis of cancer
* history of an eating disorder such as bulimia or anorexia nervosa
* surgery in the past 3 months
* surgery planned in the ensuing 6 months
* any chronic illness that could affect weight status

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2009-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in age and gender adjusted BMI z-score | 6 months

SECONDARY OUTCOMES:
Change in age and gender adjusted waist circumference percentile | 6 months
Change in age and gender adjusted blood pressure percentile | 6 months
Change in fasting lipid profile | 6 months
Change in fasting insulin and fasting glucose | 6 months
Change in plasma visfatin level | 6 months
Change in plasma adiponectin level | 6 months
Proportion of children achieving a BMI below the 85th percentile for age and gender | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Ho, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Pedersen SD, Kang J, Kline GA. Portion control plate for weight loss in obese patients with type 2 diabetes mellitus: a controlled clinical trial. Arch Intern Med. 2007 Jun 25;167(12):1277-83. doi: 10.1001/archinte.167.12.1277. PMID 17592101